CLINICAL TRIAL: NCT02356302
Title: Phase 1 Safety and Pharmacokinetics Study of MK-2048/Vicriviroc (MK-4176)/MK-2048A Intravaginal Rings
Brief Title: Safety and Pharmacokinetics of Intravaginal Rings Containing Vicriviroc (MK-4176) and/or MK-2048
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MTN-027; 12014 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2016-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vicriviroc (MK-4176) Intravaginal Ring (IVR) (Experimental): The vicriviroc (MK-4176) IVR will be inserted during the enrollment visit (Day 0), and it will be removed on Day 28.
  Interventions: Device: Vicriviroc (MK-4176) Intravaginal Ring (IVR)
- MK-2048 IVR (Experimental): The MK-2048 IVR will be inserted during the enrollment visit (Day 0), and it will be removed on Day 28.
  Interventions: Device: MK-2048 IVR
- MK-2048A IVR (Experimental): The MK-2048A IVR will be inserted during the enrollment visit (Day 0), and it will be removed on Day 28.
  Interventions: Device: MK-2048A IVR
- Placebo IVR (Placebo Comparator): The placebo IVR will be inserted during the enrollment visit (Day 0), and it will be removed on Day 28.
  Interventions: Device: Placebo IVR

INTERVENTIONS:
Device: Vicriviroc (MK-4176) Intravaginal Ring (IVR) — Contains 182 mg vicriviroc (MK-4176).
  Arms: Vicriviroc (MK-4176) Intravaginal Ring (IVR)
Device: MK-2048 IVR — Contains 30 mg MK-2048.
  Arms: MK-2048 IVR
Device: MK-2048A IVR — Contains 182 mg vicriviroc (MK-4176) and 30 mg MK-2048.
  Arms: MK-2048A IVR
Device: Placebo IVR
  Arms: Placebo IVR

SUMMARY:
Research is currently underway to develop new HIV prevention strategies. Intravaginal rings (IVRs) are one drug delivery method that is currently being studied. This study will evaluate the safety and pharmacokinetics of IVRs containing vicriviroc, MK-2048, and a combination of vicriviroc/MK-2048, in healthy, HIV-uninfected women.

DETAILED DESCRIPTION:
The development of safe and effective HIV prevention strategies is an important global health priority. IVRs have previously been approved as a delivery method for various medications, and this study will evaluate IVRs containing HIV antiretroviral medications. The purpose of this study is to assess the safety and pharmacokinetics of a combination IVR called MK-2048A that contains vicriviroc (MK-4176) and MK-2048, compared to IVRs containing vicriviroc alone and MK-2048 alone.

This study will enroll healthy, HIV-uninfected women, 18 to 45 years old. Participants will be randomly assigned to receive an IVR containing either vicriviroc, MK-2048, MK-2048A (which contains vicriviroc and MK-2048), or placebo. Participants will receive their assigned IVR at the enrollment visit, and the IVR will be removed on Day 28. Participants will attend study visits at screening, enrollment (Day 0), and Days 1, 2, 3, 7, 14, 21, 28, 29, 30, 31, and 35. Study visits may include behavioral assessments, adherence counseling and assessments, medical history reviews, physical examinations, urine collection, blood collection, pelvic specimen collection, and rectal specimen collection (optional).

ELIGIBILITY:
Inclusion Criteria:

* Born female. Note: Participants who were female at birth, who now identify as male, will not be excluded so long as they are not on female-to-male transition therapy.
* Age 18 through 45 years (inclusive) at Screening, verified per site SOPs
* Able and willing to provide written informed consent to be screened for and take part in this study (MTN-027)
* Able and willing to provide adequate locator information, as defined by the site SOPs
* HIV-uninfected, based on testing performed by study staff at Screening and Enrollment (per applicable algorithm in Appendix II of the protocol) and willing to receive results
* In general good health at Screening and Enrollment, as determined by the site Investigator of Record (IoR) or designee
* At Screening, participant states willingness to abstain from receptive sexual activity (including penile-vaginal intercourse, anal intercourse, receptive oral intercourse, finger stimulation, and the use of sex toys) for the 5 days prior to the Enrollment Visit and for the duration of study participation
* Per participant report, using an effective method of contraception at Enrollment, and intending to continue the use of an effective method for the duration of study participation. Effective methods for MTN-027 include: hormonal methods (except contraceptive IVRs), intrauterine device (IUD) inserted at least 28 days prior to enrollment, engages in sex exclusively with women, sterilized (self or partner), and/or sexually abstinent for the past 90 days.
* Women over the age of 21 (inclusive) must have documentation of a satisfactory Pap within the past 3 years prior to Enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009), or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result
* Per participant report at Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, or vaginal products for the duration of study participation
* Per participant report at Screening, regular menstrual cycles with at least 21 days between menses. Note: This criterion is not applicable to participants who report using a progestin-only method of contraception at Screening, e.g., Depo-Provera or levonorgestrel-releasing IUD nor to participants using continuous combination oral contraceptive pills, as the absence of regular menstrual cycles is an expected, normal consequence in this context.
* At Screening, participant states a willingness to refrain from inserting any non-study vaginal products or objects into the vagina, including, but not limited to, spermicides, female condoms, diaphragms, contraceptive IVRs, vaginal medications, menstrual cups, cervical caps (or any other vaginal barrier method), douches, lubricants, sex toys (vibrators, dildos, etc.) for the 5 days prior to Enrollment and for the duration of their study participation

Exclusion Criteria:

* Participant report of any of the following at Screening and/or Enrollment:

  * History of adverse reactions to any of the components of the study products
  * Non-therapeutic injection drug use in the 12 months prior to Screening and Enrollment
  * Post-exposure prophylaxis (PEP) for HIV exposure within 6 months prior to Enrollment
  * Pre-exposure prophylaxis (PrEP) for HIV prevention within the 6 months prior to Enrollment
  * Regular use and/or anticipated regular use during the period of study participation of CYP3A inducer(s) and/or inhibitor(s)
  * Use and/or anticipated use during the period of study participation of female-to-male transition therapy
  * Chronic and/or recurrent candidiasis
  * Gonorrhea, chlamydia, and/or syphilis diagnosis in the 6 months prior to Enrollment
  * Last pregnancy outcome 90 days or less prior to Screening
  * Currently breastfeeding
  * Has had a hysterectomy
  * Intends to become pregnant within the next 3 months
  * Has plans to relocate away from the study site area in the next 3 months
  * Current sexual partner is known to be HIV-positive
* Reports participating in any other research study involving drugs, medical devices, or vaginal products within 60 days or less prior to enrollment
* At Screening or Enrollment, as determined by the IoR/designee, any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease
* Has any of the following laboratory abnormalities at Screening:

  * Aspartate aminotransferase (AST) or alanine transaminase (ALT) Grade 1 or higher
  * Calculated creatinine clearance less than 60 mL/min by the Cockcroft-Gault formula, where creatinine clearance (female) in mL/min = (140 - age in years) x (weight in kg) x (0.85)/72 x (creatinine in mg/dL)
  * Hemoglobin Grade 1 or higher
  * Platelet count Grade 1 or higher
  * White blood count Grade 2 or higher
  * Positive HBsAg test result
  * Positive anti-hepatitis C virus (HCV) test result
  * International normalized ratio (INR) greater than 1.5 × the site laboratory upper limit of normal (ULN)
  * Note: Otherwise eligible participants with an exclusionary test result (other than HIV, hepatitis B virus [HBV], or HCV) can be re-tested during the screening process. If a participant is re-tested and a non-exclusionary result is documented within 45 days of providing informed consent for screening, the participant may be enrolled.
* Pregnant at either Screening or Enrollment. Note: A documented negative pregnancy test performed by study staff is required for inclusion; however a self-reported pregnancy is adequate for exclusion from screening/enrollment into the study.
* Diagnosed with urinary tract infection (UTI) at Screening or Enrollment. Note: Otherwise eligible participants diagnosed with UTI during screening will be offered treatment. If within the 45 day screening window treatment is complete and symptoms have resolved the participant may be enrolled.
* Diagnosed with pelvic inflammatory disease, reproductive tract infection (RTI) or a sexually transmitted infection (STI) requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines (http://www.cdc.gov/std/treatment/) at Screening or Enrollment. Note: With the exception of gonorrhea, chlamydia, and/or syphilis, otherwise eligible participants diagnosed with a RTI during screening will be offered treatment. If within the 45 day screening window treatment is complete and symptoms have resolved the participant may be enrolled.
* At Enrollment, has a clinically apparent Grade 1 or higher pelvic exam finding (observed by study clinician or designee) per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009), Addendum 1, Female Genital Grading Table for Use in Microbicide Studies. Note: Cervical friability bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the IoR/designee is considered expected non-menstrual bleeding and is not exclusionary.
* At Screening, severe pelvic relaxation such that either the vaginal walls or the uterine cervix descend beyond the vaginal introitus with valsalva maneuver or has pelvic anatomy that compromises the ability to adequately assess vaginal safety
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Proportion of women in each of the four IVR regimens with genitourinary events Grade 1 or higher judged to be related to study product | Measured through Day 35
  As defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Dec 2004 (Clarification dated August 2009), Addendum 1, (Female Genital Grading Table for Use in Microbicide Studies)
Proportion of women in each of the four IVR regimens with adverse events Grade 2 or higher | Measured through Day 35
  As defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Dec 2004 (Clarification dated August 2009)
Measurement of local and systemic concentrations of vicriviroc (MK-4176) | Measured through Day 35
  In plasma, vaginal fluids, and cervical tissue during and after 28 days of continuous use of an IVR containing 182 mg vicriviroc (MK-4176), or 30 mg MK-2048, or 182 mg vicriviroc (MK-4176) + 30 mg MK-2048 (MK-2048A)
Measurement of local and systemic concentrations of MK-2048 | Measured through Day 35
  In plasma, vaginal fluids, and cervical tissue during and after 28 days of continuous use of an IVR containing 182 mg vicriviroc (MK-4176), or 30 mg MK-2048, or 182 mg vicriviroc (MK-4176) + 30 mg MK-2048 (MK-2048A)

SECONDARY OUTCOMES:
Participant report of acceptability | Measured through Day 35
  Including genitourinary and emotional (dis)comfort, awareness/feeling during daily activities, ring insertion/removal issues, and willingness to use in the future
Participant report of frequency of study IVR removal/expulsion and duration without IVR inserted in vagina | Measured through Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hoesley, MD, Study Chair — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - Alabama CRS, Birmingham, Alabama
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Hoesley CJ, Chen BA, Anderson PL, Dezzutti CS, Strizki J, Sprinkle C, Heard F, Bauermeister J, Hall W, Jacobson C, Berthiaume J, Mayo A, Gundacker H, Richardson-Harman N, Piper J; Microbicide Trials Network 027 Study Team. Phase 1 Safety and Pharmacokinetics Study of MK-2048/Vicriviroc (MK-4176)/MK-2048A Intravaginal Rings. Clin Infect Dis. 2019 Mar 19;68(7):1136-1143. doi: 10.1093/cid/ciy653. PMID 30289435